CLINICAL TRIAL: NCT04037553
Title: The Changes of Endotracheal Tube Cuff Pressures After Ear, Head and Neck Surgery-Related Positions: A Prospective Observational Study
Brief Title: Changes of Endotracheal Tube Cuff Pressures After Ear, Head and Neck Surgery Positions
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, Associate Professor, Istanbul University
Other Study IDs: 2019/156
Record Dates: First submitted 2019-07-03; First posted 2019-07-30 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Endotracheal Tube Cuff Pressure; Surgery; Ear; Surgery; Head and Neck; Position
Keywords: Endotracheal tube cuff pressure; Ear Surgery; Head and Neck Surgery; Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Patients underwent right ear surgery: After intracuff pressure (ICP) is adjusted to 25 cmH2O at neutral position, lateral neck rotation (approximately 60-70 degrees to the left) was applied to the patients and ICP values were documented following 3 respiration cycles.
  Interventions: Other: Intracuff pressure measurement
- Group 2: Patients underwent left ear surgery: After intracuff pressure (ICP) is adjusted to 25 cmH2O at neutral position, lateral neck rotation (approximately 60-70 degrees to the right) was applied to the patients and ICP values were documented following 3 respiration cycles.
  Interventions: Other: Intracuff pressure measurement
- Group 3: Patients underwent left head and neck surgery: After intracuff pressure (ICP) is adjusted to 25 cmH2O at neutral position, gel pillow with the height of 4,5 cm was placed under the shoulders of patients to extend the neck. Following 3 respiration cycles, the ICPs were noted. Then, right or left lateral neck rotation was applied depending on the operation side (approximately 60-70 degree to the opposite site). After 3 respiration cycles, ICPs were documented again.
  Interventions: Other: Intracuff pressure measurement

INTERVENTIONS:
Other: Intracuff pressure measurement — Intracuff pressure values were monitorized and noted before and after head and neck positions and during the surgeries at 15th, 30th, 60th and 90th minutes at related positions and just before extubation at neutral position.
  Groups: Group 1
Other: Intracuff pressure measurement — Intracuff pressure values were monitorized and noted before and after head and neck positions and during the surgeries at 15th, 30th, 60th and 90th minutes at related positions and just before extubation at neutral position.
  Groups: Group 2
Other: Intracuff pressure measurement — Intracuff pressure values were monitorized and noted before and after head and neck positions and during the surgeries at 15th, 30th, 60th and 90th minutes at related positions and just before extubation at neutral position.
  Groups: Group 3

SUMMARY:
Increased or decreased intracuff pressures (ICPs) of cuffed endotracheal tubes (cETTs) can lead to many morbidities.The ICPs of cETTs can be changed by the the patients' ear and head&neck surgery positions. We performed this study to show the effect of the routine combination of neck positions on ICP whilst ear and head& neck surgeries.

A total of 90 patients were enrolled to the study. Groups 1 and 2 included the patients who underwent right and left ear surgeries, respectively. Group 3 included all patients undergoing head and neck surgery.After the general anesthesia induction, the patients were given a neutral position.The first ICP was measured and adjusted to 18,4 mm Hg (25 cmH2O) at neutral position. Left or right neck rotation was applied to Group 1 or 2 in conformity with the ear operation site and ICP value was documented. Gel pillow with the height of 4,5 cm was placed under the shoulders of Group 3 patients to extend the neck and the ICP was noted. Then, right or left neck rotation was applied depending on the operation side and ICP was documented again. Additionally, ICP values were monitorized continuously in all patients during the surgeries, and documented at 15th, 30th, 60th and 90th minutes at related positions and just before extubation at neutral position. If the ICP value fell below 14,7 mmHg (20 cmH2O) or rose above 22 mmHg (30 cmH2O), ICP was adjusted to 18,4 mm Hg (25 cmH2O) again.

DETAILED DESCRIPTION:
Increased or decreased intracuff pressures (ICPs) of cuffed endotracheal tubes (cETTs) can lead to many morbidities. Guidelines recommend that the ICP should be kept between 20 and 30 cmH2O. Over inflation of the cuff can cause tracheal mucosal injury ,tracheal stenosis, tracheoesophageal fistula, postoperative stridor, laryngospasm, laryngeal nerve damage and tracheal rupture. However, under inflation can cause air leakage, aspiration and ventilation associated pneumonia.The cETT can be displaced by movement of the patients' heads and necks while positioning for surgeries of ear, head and neck. These positionings and displacements may be the reasons of changes in ICPs. The investigators performed this study to show the effect of the routine combination of neck positions on ICP whilst ear, head and neck surgeries.

After obtaining ethics committee approval and written informed consent, 90 patients with American Society of Anesthesiologists (ASA) physical status I-III and aged older than 18 years were enrolled to the study. The patients were allocated to 3 groups according to their surgery types. Groups 1 and 2 included the patients who underwent right and left ear surgeries, respectively. Group 3 included all patients undergoing head and neck surgery without considering the surgical site. After the general anesthesia induction, the patients were given a neutral position defined by Komasawa et al. The first ICP was measured and adjusted to 18,4 mm Hg (25 cmH2O) at neutral position just after taping the tube and monitoring the 3 consecutive respiration cycles. After neutral measurements, left or right neck rotation (approximately 60-70 degree to the opposite site) was applied to Group 1 or 2 in conformity with the ear operation site and ICP value was documented following 3 respiration cycles. Gel pillow with the height of 4,5 cm was placed under the shoulders of Group 3 patients to extend the neck. After waiting for 3 respiration cycles, the ICP was noted. Then, right or left neck rotation was applied depending on the operation site (approximately 60-70 degree to the opposite site). Following 3 respiration cycles, ICP was documented again. Additionally, ICP values were monitorized continuously in all patients during the surgeries, and documented at 15th, 30th, 60th and 90th minutes at related positions and just before extubation at neutral position. At any time point, if ICP value fell below 14,7 mmHg (20 cmH2O) or rose above 22 mmHg (30 cmH2O), ICP was adjusted to 18,4 mm Hg (25 cmH2O) again. After all data were collected, statistical analysis were performed by using Statistical Package for the Social Sciences (SPSS) version 22.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* American Society of Anesthesiologists (ASA) physical status I-III
* Patients who scheduled for elective ear or head and neck surgery under general anesthesia

Exclusion Criteria:

* Morbid obesity (body mass index (BMI) >35)
* Limited neck movements
* Previous history of radiotherapy or surgery to the head and neck area
* Nasotracheal intubation under general anesthesia
* Peroperative tracheotomy requirements
* Respiratory tract infection
* Surgery planned for midline neck masses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective ear or head and neck surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Intracuff Pressure | 0th minute (just after the positioning from neutral to surgical position)
  Endotracheal Tube Cuff Pressures After Ear, Head and Neck Surgery Positions

SECONDARY OUTCOMES:
Intracuff Pressure | 15th minute
  Endotracheal Tube Cuff Pressure at 15th minute at surgery-related position
Intracuff Pressure | 30th minute
  Endotracheal Tube Cuff Pressure at 30th min at surgery-related position
Intracuff Pressure | 60th minute
  Endotracheal Tube Cuff Pressure at 60th min at surgery-related position
Intracuff Pressure | 90th minute
  Endotracheal Tube Cuff Pressure at 90th min at surgery-related position
Intracuff Pressure | At the end of the surgery before extubation
  Endotracheal Tube Cuff Pressure just before extubation at neutral position

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salviz, MD, Principal Investigator — MD, Assoc.Prof.
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Result] Lizy C, Swinnen W, Labeau S, Poelaert J, Vogelaers D, Vandewoude K, Dulhunty J, Blot S. Cuff pressure of endotracheal tubes after changes in body position in critically ill patients treated with mechanical ventilation. Am J Crit Care. 2014 Jan;23(1):e1-8. doi: 10.4037/ajcc2014489. PMID 24382623
- [Result] Komasawa N, Mihara R, Imagawa K, Hattori K, Minami T. Comparison of Pressure Changes by Head and Neck Position between High-Volume Low-Pressure and Taper-Shaped Cuffs: A Randomized Controlled Trial. Biomed Res Int. 2015;2015:386080. doi: 10.1155/2015/386080. Epub 2015 Oct 5. PMID 26509152